CLINICAL TRIAL: NCT06994247
Title: Impact of Phenotypic and Psychological Characteristics and a Motivational Telephone Intervention on Continuous Positive Airway Pressure (CPAP) Adherence in Patients With Severe Obstructive Sleep Apnea
Brief Title: Boosting CPAP Use in Adults With Severe Sleep Apnea: Role of Motivation and Psychological Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2181-198-03-04-24-0107
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Telephone Call - Intervention Group (Experimental): Participants in this group will receive standard CPAP therapy along with a motivational telephone intervention. Approximately one month after initiating CPAP therapy, a physician will contact participants by phone to assess usage and discuss any difficulties. During the call, the physician will provide personalized motivation and education regarding the health benefits of consistent CPAP use to enhance treatment adherence.
  Timing: At 1 month post-enrollment Delivered by: Medical doctor Mode: Telephone Goal: To improve CPAP adherence at the 3-month follow-up
  Interventions: Behavioral: Motivational Telephone Call
- No Intervention - Control Group (No Intervention): Participants in this group will receive standard CPAP therapy only, without any additional motivational contact beyond routine clinical follow-up. Data on adherence will be collected at the 3-month time point using CPAP device memory cards.

INTERVENTIONS:
Behavioral: Motivational Telephone Call — This intervention consists of a single, personalized motivational telephone call delivered by a medical doctor, one month after initiation of CPAP treatment, uniquely timed to address early barriers and enhance self-efficacy. Unlike standard care or automated follow-ups, it offers tailored support based on patient experience, making it a low-cost yet targeted behavioral strategy to improve adherence. Content of the telephone call includes inquiry about patient's experience with CPAP therapy, identification of barriers to regular use, education on the health benefits of consistent CPAP usage, and personalized motivational messages aimed at increasing compliance.
  Arms: Motivational Telephone Call - Intervention Group

SUMMARY:
The goal of this randomized prospective clinical trial is to examine whether phenotypic traits, psychological characteristics, assessed by STAI (engl. The State-Trait Anxiety Inventory) and IPIP50S (engl. International Personality Item Pool) questionnaires, and patients' self-efficacy, assessed by SEMSA (engl. Self-Eficacy Measure for Sleep Apnea) questionnaire, are associated with CPAP adherence after three months of use. The study also evaluates whether a motivational phone call one month after therapy initiation improves CPAP adherence at the three-month follow-up. The main questions it aims to answer are:

* Are phenotypic and psychological traits associated with adherence to CPAP therapy after 3 months of treatment?
* Can a single motivational telephone intervention, one month after initiating CPAP therapy, significantly improve CPAP adherence at the three-month follow-up compared to no intervention? Researchers will compare patients who receive a phone call to those who do not, to see if this simple intervention leads to better CPAP adherence after three months of use.

Participants will:

* Undergo polysomnography before starting CPAP therapy,
* Complete three questionnaires (IPIP50S, STAI, SEMSA) before starting CPAP therapy,
* Be randomly assigned to either receive a motivational phone call one month after starting CPAP therapy or to a control group without any phone call,
* Be invited for a follow-up after three months of CPAP use to download and analyze CPAP adherence data from their CPAP devices.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older
* Diagnosis of severe obstructive sleep apnea (OSA), defined as AHI ≥30
* Signed informed consent for participation in the study
* Adequate physical and psychological capacity to participate in the intervention and complete questionnaires
* Patients who are initiating CPAP therapy at the Sleep Medicine Center, University of Split School of Medicine
* Availability for follow-up over a three-month period

Exclusion Criteria:

* Presence of central sleep apnea or other primary sleep disorders
* Cognitive impairment or psychiatric conditions that may hinder the ability to follow instructions or complete questionnaires
* Previous experience with CPAP therapy prior to study enrollment
* Significant comorbidities (e.g. unstable cardiovascular disease, advanced pulmonary disease) that may interfere with study outcomes
* Pregnancy
* Inability to participate in follow-up assessments or be contacted by telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
CPAP Adherence After Three Months of Therapy | From baseline (enrollment) to 3-month follow-up
  CPAP adherence at three months, measured as the percentage of days with CPAP usage ≥4 hours per night, obtained from CPAP device memory cards.

SECONDARY OUTCOMES:
Baseline self-efficacy related to OSA treatment | Baseline
  Self-efficacy related to obstructive sleep apnea (OSA) treatment will be assessed at baseline using the Self-Efficacy Measure for Sleep Apnea (SEMSA) questionnaire. The SEMSA is a validated self-report instrument with scores ranging from 1 to 4, where higher scores indicate greater self-efficacy (i.e., more confidence in using CPAP). The total score is continuous and will be analyzed as a predictor of CPAP adherence at 3 months.
Baseline anxiety levels (state and trait) | Baseline
  Anxiety levels will be assessed at baseline using the State-Trait Anxiety Inventory (STAI), a validated self-report instrument consisting of two subscales: state anxiety and trait anxiety. Each subscale yields a score from 20 to 80, with higher scores indicating greater anxiety. Both scores will be analyzed separately as continuous predictors of CPAP adherence at 3 months.
Baseline personality traits | Baseline
  Personality traits will be measured at baseline using the International Personality Item Pool - 50-item Short Form (IPIP-50). The IPIP-50 evaluates five personality traits: Openness, Conscientiousness, Extraversion, Agreeableness, and Neuroticism. Each trait score is derived from responses on a 1 to 5 Likert scale, with higher scores indicating a stronger presence of that trait. Each trait will be analyzed separately as a categorical or continuous predictor of CPAP adherence at 3 months.
Effect of motivational telephone intervention | From baseline to 3-month follow-up
  Binary exposure variable (intervention: yes/no). CPAP adherence at 3 months will be compared between the intervention and control groups to assess the effect of the motivational telephone intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Split School of Medicine, Split, Dalmatia, Croatia

IPD SHARING:
Plan to Share IPD: No